CLINICAL TRIAL: NCT06815900
Title: Correlation Between Sleep Quality , Physical Fitness and Body Mass Index in Physical Therapy Students
Brief Title: Correlation Between Sleep Quality , Physical Fitness and Body Mass Index
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Toka Ahmed Fayez Mohamed, researcher physiotherapist, Cairo University
Other Study IDs: P.T.REC/012/005496
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Sleep Quality , Physical Fitness and Body Mass Index
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- one group: observational study of this group
  Interventions: Other: one group .observational study

INTERVENTIONS:
Other: one group .observational study — observational study of this group

SUMMARY:
It is estimated that 10-13% of adults suffer from chronic insomnia. Short sleep duration is linked to obesity, type 2 diabetes, high blood pressure, and cardiovascular diseases. Feeling tired during the day predicts poor sleep quality (SQ), while wakefulness is linked to better SQ. Previous studies have also reported a relationship between short sleep duration and increased Body Mass Index (BMI), and a high correlation between increased BMI and decreased SQ, with more frequent awakenings. Moreover, there is a connection between sleep disorders and weight gain. The study is significant because it aims to uncover the relationships between sleep quality, physical fitness, and body mass index (BMI) in physical therapy students, offering insights crucial for improving their health and academic performance. By identifying how these factors interact, the study can inform targeted interventions to enhance student well-being, clinical competence, and long-term health. Additionally, the findings can guide educational programs to support healthier lifestyles and enable students to serve as effective role models for their future patients, thereby contributing to overall healthcare quality.

ELIGIBILITY:
Inclusion Criteria:

* Student of both gender with age that ranges from 18 to 25 years old.
* Must be actively enrolled in an accredited physical therapy program.
* Open to students from any year of study within the physical therapy program.

Exclusion Criteria:

* Diagnosed with sleep disorders such as insomnia, sleep apnea, or narcolepsy.
* Chronic physical conditions like cardiovascular, respiratory, neurological, or musculoskeletal disorders.
* Metabolic or endocrine disorders such as diabetes or thyroid disorders.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: both male and female aged between 18-25 years old
Sampling Method: Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
sleep quality | six months
  questionnaire
physical fitness | six months
  questionnaire
body mass index | six months
  body mass index international equation

IPD SHARING:
Plan to Share IPD: Undecided